CLINICAL TRIAL: NCT05684211
Title: A Multicenter, Open-label, Parallel-group，Randomised, Phase IIb Trial of Efficacy and Safety of Ametumumab in Combination With Anti-PD-1 Monoclonal Antibody and FOLFIRI Versus Ametumumab or Cetuximab in Combination With FOLFIRI in Patients With RAS Wild-type Advanced Colorectal Cancer
Brief Title: A Study of Ametumumab in Combination With Anti-PD-1 Monoclonal Antibody and FOLFIRI in Patients With RAS Wild-type Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Celfuture Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WBP252-004
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — spartalizumab; Cetuximab; IFL protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ametumumab (QW) + anti-PD-1 monoclonal antibody+ FOLFIRI (Active Comparator): Ametumumab 450 mg/m2 (QW) + anti-PD-1 monoclonal antibody (in the case of toripalimab 3 mg/kg, Q2W) + FOLFIRI;
  Interventions: Drug: Ametumumab; Drug: Anti-PD-1 monoclonal antibody; Drug: FOLFIRI
- Ametumumab(Q2W) + anti-PD-1 monoclonal antibody + FOLFIRI; (Active Comparator): Ametumumab 450 mg/m2 (Q2W) + anti-PD-1 monoclonal antibody (in the case of toripalimab 3 mg/kg, Q2W) + FOLFIRI;
  Interventions: Drug: Ametumumab; Drug: Anti-PD-1 monoclonal antibody; Drug: FOLFIRI
- Ametumumab (Q2W) + FOLFIRI; (Active Comparator): Ametumumab 450 mg/m2 (Q2W) + FOLFIRI
  Interventions: Drug: Ametumumab; Drug: FOLFIRI
- Cetuximab + FOLFIRI; (Active Comparator): Cetuximab 500 mg/m2 (Q2W) + FOLFIRI
  Interventions: Drug: Cetuximab; Drug: FOLFIRI

INTERVENTIONS:
Drug: Ametumumab — A recombinant fully human anti-EGFR monoclonal antibody
  Arms: Ametumumab (Q2W) + FOLFIRI;; Ametumumab (QW) + anti-PD-1 monoclonal antibody+ FOLFIRI; Ametumumab(Q2W) + anti-PD-1 monoclonal antibody + FOLFIRI;
Drug: Anti-PD-1 monoclonal antibody — Toripalimab 3 mg/kg，Intravenous titration，Q2W
  Arms: Ametumumab (QW) + anti-PD-1 monoclonal antibody+ FOLFIRI; Ametumumab(Q2W) + anti-PD-1 monoclonal antibody + FOLFIRI;
Drug: Cetuximab — Cetuximab 500 mg/m2 ，Intravenous titration，Q2W
  Arms: Cetuximab + FOLFIRI;
Drug: FOLFIRI — Rinotecan hydrochloride，180mg/m2，intravenous titration，Q2W； 5 -Fluorouracil，400 mg/ m2, intravenous push, then 1200 mg/ m2 /day x 2 days, intravenous titration,Q2W; Calcium folinate,400mg/m2,intravenous titration，Q2W

SUMMARY:
This is a multicenter, open-label, parallel-group, randomised, A phase IIb clinical trial of efficacy and safety of Ametumumab in combination with anti-PD-1 monoclonal antibody and FOLFIRI versus Ametumumab or Cetuximab in combination with FOLFIRI in patients with RAS wild-type advanced colorectal cancer.

DETAILED DESCRIPTION:
This is a multicenter, open-label, parallel-group, randomised, phase IIb trial. This study is to evaluate and compare the efficacy and safety of Ametumumab (anti-EGFR monoclonal antibody) combined with anti-PD-1 monoclonal antibody in first-line treatment of RAS wild-type colorectal cancer patients, as well as to assess the immunogenicity and pharmacokinetic profile and recommend dosing regimen for phase III clinical trials.Conditions and keywords.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily sign written informed consent; Age 18 ~ 85 years (inclusive), male or female;

•Patients requiring first-line treatment for locally advanced colorectal cancer with distant metastasis or unresectable disease; Histologically or cytologically confirmed adenocarcinoma of the colon or rectum; RAS (KRAS, NRAS) gene is wild-type and no BRAF V600E mutation has been identified; Presence of at least one measurable lesion (non-radiation field) confirmed by CT or MRI that meets RECIST 1.1 criteria; Performance status (ECOG) score 0 or 1.

Exclusion Criteria:

Previous chemotherapy for colorectal cancerPrevious treatment with anti-EGFR monoclonal antibodies Received systemic anti-tumor treatment approved or of other clinical studies within 4 weeks prior to the first dose.

Radiotherapy or surgery within 4 weeks prior to enrollment, except for diagnostic biopsy Participation in other clinical trials within 4 weeks prior to enrollment; Severe skin disease requiring systemic treatment. Presence of serious clinical infection.\ Uncontrolled pleural effusion, pericardial effusion or peritoneal effusion after treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | PFS will be measured from the date of first dose of study drug until first documented clinical or radiographic evidence of disease progression by RECIST 1.1, clinical progression, start of new therapy or death. approximately 45 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | ORR is defined as a CR or PR per RECIST version 1.1 recorded from the date of randomization until date of first documentation of PD, death, or start of new anti-cancer therapy, approximately 45 months.
incidence of adverse events | Incidence and severity of AEs graded according to the NCI CTCAE v5.0, Duration of study, approximately 45 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China